CLINICAL TRIAL: NCT03211936
Title: Pulmonary Evaluation at Different Levels of PEEP: Ultrasonography Compared to Electrical Impedance Tomography (TIE) During Intraoperative Elective Surgeries
Brief Title: Pulmonary Evaluation With Ultrasound in Different Levels of PEEP
Acronym: EVALUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NP 807/15
Record Dates: First submitted 2017-04-20; First posted 2017-07-11 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Atelectasis; Hypertension; Lung Edema
MeSH Terms: conditions — Pulmonary Atelectasis; Hypertension; Pulmonary Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP 4 (Active Comparator): We titrate peep, using tomography impedance, making ultrasound after "level by level' of peep. After titrated peep we setup peep 4 and maintained during the procedure.
  * PEEP 4 cmH2O
  * Use ultrasound
  Interventions: Procedure: PEEP TITRATED; Device: Use ultrasound; Device: Impedance tomography; Other: PEEP 4
- PEEP TITRATED (Experimental): We titrate peep, using tomography impedance, making ultrasound after "level by level' of peep. After tritiated peep we setup the best peep for less collapse (using the tomography of electrical impedance) and maintained during the procedure.
  * PEEP titrated
  * Use ultrasound
  * Impedance tomography
  * Best PEEP for less collapse
  Interventions: Procedure: PEEP TITRATED; Device: Use ultrasound; Device: Impedance tomography; Other: Best PEEP for less collapse

INTERVENTIONS:
Procedure: PEEP TITRATED — After titrated peep levels, we choice this level of peep for de group (peep titrated)
Device: Use ultrasound — We make a lung ultrasound after we setup a different level of PEEP
Device: Impedance tomography — We use the impedance tomography to titrate peep levels, and acquire dates of collapse, hyperdistension and compliance.
Other: Best PEEP for less collapse — After titrated PEEP levels we setup the best PEEP the according of tomography impedance
  Arms: PEEP TITRATED
Other: PEEP 4 — We set the peep level after titrated peep = 4 cmH20.
  Arms: PEEP 4

SUMMARY:
Patients submitted to general anesthesia and artificial ventilation almost always develop pulmonary atelectasis, which can determine adverse consequences both intraoperatively and postoperatively. It is recommended to use physiological tidal volume (6 - 8 mL / kg of ideal body weight) during the intraoperative period in order to minimize the risk of lung injury. To prevent the formation of atelectasis, minimizing the risk of complications, the use of PEEP has been recommended. At present, there is no way to make an optimal adjustment of PEEP to the needs of each patient, seeking a value that keeps the alveoli open without forming atelectasis and also without areas of hyperdistension.

The aim of this study was to evaluate the agreement between the ultrasound and the electrical impedance tomography - Timpel® (TIE) to detect the beginning of the formation of areas of atelectasis after pulmonary recruitment, with decreasing PEEP values. In addition, the lung ultrasound will be validated for intraoperative use for both adequacy of PEEP, as well as quantitative analyzes of ultrasound images to assess atelectasis.

18 patients (> 18 years) of both sexes, submitted to general anesthesia, will be prospectively studied. All patients will receive, in addition to the usual monitoring, the monitoring with the electrical impedance tomography and chest ultrasonography, after being anesthetized and under neuromuscular block, being ventilated with an inspired fraction of 50% oxygen (or greater to maintain oxygen saturation > 96% ), Tidal volume of 6 mL / kg and respiratory rate to maintain expiratory tidal CO2 between 35-45 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and female patients, over 18 years of age, who undergo abdominal surgeries (prostatectomies and hysterectomies) and who do not have preexisting pulmonary diseases. They will be approached in the room prior to surgery, at which time the purpose of the research will be explained, besides making clear that it will not entail costs and so little any injury, scar, or damage. If accepted by the patient, the consent form will be applied.

Exclusion Criteria:

* Exclusion criteria for the study will be: patients classified by the American Society of Anesthesiologists Physical status as ASA-3 or above, patients with obstructive and restrictive respiratory diseases, patients with predictable orotracheal intubation difficulties (eg, obese patients) who require Manipulation of the upper airways. Also excluded are patients with pacemakers and patients scheduled for procedures in the thoracic region

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Hyperdistension | during tritiate peep
  We acquire lung ultrasound images during tritiating peep and analyze if any patient have hyperdistension

SECONDARY OUTCOMES:
Atelectasis | in the final of the procedure
  After the procedure we analyze with patient group have more atelectasis

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Carmona, PhD, Study Chair — University of Sao Paulo; Claudia Simões, PhD, Study Director — Universiadde de São Paulo/ ICESP

IPD SHARING:
Plan to Share IPD: No